CLINICAL TRIAL: NCT02463812
Title: Energy Supplement With Lipid Emulsion Following Major Surgery
Brief Title: Lipid Infusion Following Major Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00055553
Record Dates: First submitted 2015-04-21; First posted 2015-06-04 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2016-10

CONDITIONS: Parenteral Nutrition
MeSH Terms: conditions — Hyperphagia | interventions — soybean oil, phospholipid emulsion; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intralipid (Experimental): Patients will receive Intralipid infusion in the recovery room.
  Interventions: Drug: Intralipid
- Control (Placebo Comparator): Patients will receive infusion of normal saline in the recovery room.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Intralipid
  Arms: Intralipid
Drug: Saline
  Arms: Control

SUMMARY:
Surgery puts a lot of stress on the body, and during recovery from surgery, the body uses a lot of energy to help with healing and getting stronger. Often, sugars are given before surgery to help give the body an energy boost. Lipid solutions can also be used as an energy source and are commonly used as supplements in patients needing long-term nutrition from an intravenous route (e.g., total parenteral nutrition) when they can not eat by mouth for a medical reason. Intralipid, a solution of lipid molecules from soybeans and eggs, is commonly used for patients who need nutrition and energy supplements. The investigators wish to test whether giving Intralipid immediately after surgery can improve recovery from major surgery.

DETAILED DESCRIPTION:
BACKGROUND The perioperative events associated with major surgery trigger the body's stress response, compromising optimal post-surgical recovery and outcomes. Moreover, traditional perioperative indications, such as restricting food up to two days before surgery, have been shown to be associated with poor outcomes following surgery. The Enhanced Recovery After Surgery (ERAS) protocol, initiated in the early 2000's, aimed to address these problems. The ERAS protocol has recommendations for pre-, intra-, and post-operative stages, with the goal of modifying physiological and psychological responses to surgery. A key component of ERAS is perioperative nutrition, including avoidance of fasting before surgery and carbohydrate loading up to two hours pre-surgery. It is hypothesized that adequate nutrition and provision of an energy source in the perioperative period can attenuate the body's stress response during surgery, thereby enabling faster and more successful recovery.

Early post-operative feeding is another recommendation of ERAS and is also intended to ensure optimal metabolic balance. Post-operative nutrition of ERAS patients generally involves oral feeding with energy-dense nutritional supplements in the days after surgery until the patient is ready for normal food intake. Lipids and carbohydrates form the bulk of these supplements, providing a readily available energy source. Lipid emulsions, such as Intralipid®, are used commonly in total parenteral nutrition and are also indicated as an energy source in patients for whom the usual intravenous fluid therapy would not be adequate. Lipid emulsions alone may therefore be helpful in enhancing recovery following major surgery, particularly in patients who are not good candidates for a strict ERAS protocol. With respect to short-term outcomes following surgery, Intralipid has been shown to modulate blood pressure by increasing systemic vascular resistance and cardiac output.

Only one study so far has evaluated post-surgery recovery outcomes following administration of lipid emulsion exclusively. The investigators found that patients receiving an intravenous infusion of lipid emulsion experienced better overall recovery and faster time eye opening and exit from the operating room compared to patients receiving an infusion of 0.9% normal saline. While these results suggest that post-operative lipid delivery improves recovery, the study did not assess differences in basic vital signs between the two groups, and the subjects were limited to those undergoing laparoscopic cholecystectomy. In this study, the investigators will recruit patients undergoing any surgery of the abdomen and assess post-operative outcomes, including vital signs, following an intravenous bolus of Intralipid® 20% or 0.9% normal saline.

OBJECTIVE To demonstrate that patients receiving an intravenous bolus of Intralipid® 20% immediately following surgery experience improved post-surgical recovery compared to patients receiving an intravenous saline bolus.

HYPOTHESIS The investigators hypothesize that patients who receive an intravenous bolus of Intralipid® following major abdominal surgery will show more stable vital signs and faster discharge from the recovery room compared to patients receiving a saline bolus.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* Scheduled for abdominal surgery
* Provide written, informed consent

Exclusion Criteria:

* Patient refusal
* Pre-existing neurological deficit
* Existing or potential for coagulation abnormality
* Local or systemic infection
* Allergy to local anesthetic
* Contraindication to propofol
* Liver disease/compromised liver metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure at discharge from PACU | During stay in recovery room (expected average 2 hrs)
  Overall primary outcome will be collective vital signs
Change in respiration rate at discharge from PACU | During stay in recovery room (expected average 2 hrs)
  Overall primary outcome will be collective vital signs
Change in pulse at discharge from PACU | During stay in recovery room (expected average 2 hrs)
  Overall primary outcome will be collective vital signs
Change in oxygen saturation at discharge from PACU | During stay in recovery room (expected average 2 hrs)
  Overall primary outcome will be collective vital signs

SECONDARY OUTCOMES:
Total volume of fluid required in recovery room | During stay in recovery room (expected average 2 hrs)
Total dosage of vasopressor required in recovery room | During stay in recovery room (expected average 2 hrs)
Length of stay in recovery room | Upon discharge from PACU (expected average 2 hrs post-surgery)
Length of stay in hospital | Upon discharge from hospital (expected 4-5 days post-surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Li Q, Yang D, Liu J, Zhang H, Zhang J. Intravenous lipid emulsion improves recovery time and quality from isoflurane anaesthesia: a double-blind clinical trial. Basic Clin Pharmacol Toxicol. 2014 Aug;115(2):222-8. doi: 10.1111/bcpt.12223. Epub 2014 Mar 24. PMID 24612915
- [Background] Soop M, Carlson GL, Hopkinson J, Clarke S, Thorell A, Nygren J, Ljungqvist O. Randomized clinical trial of the effects of immediate enteral nutrition on metabolic responses to major colorectal surgery in an enhanced recovery protocol. Br J Surg. 2004 Sep;91(9):1138-45. doi: 10.1002/bjs.4642. PMID 15449264
- [Background] Varadhan KK, Lobo DN, Ljungqvist O. Enhanced recovery after surgery: the future of improving surgical care. Crit Care Clin. 2010 Jul;26(3):527-47, x. doi: 10.1016/j.ccc.2010.04.003. PMID 20643305